CLINICAL TRIAL: NCT01310738
Title: Multicentric Efficacy and Safety Study of Antileishmanial Drugs for Treatment of Visceral Leishmaniasis in Brazil
Brief Title: Efficacy and Safety Study of Drugs for Treatment of Visceral Leishmaniasis in Brazil
Acronym: LVBrasil
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: DSMB recommendation based on programmed interim analysis.
Sponsor: University of Brasilia (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Drugs for Neglected Diseases (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Gustavo Adolfo Sierra Romero, Professor, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LVBrasil_2007; 559819/2010-2 (Other Grant/Funding Number: CNPq - Brazil); 108042500 (Other Grant/Funding Number: Finaciadora de Estudos e Projetos - FINEP - Brazil); CAAE 0973.1.000.245-10 (Other: Brazilian National Ethics Council)
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Visceral Leishmaniasis
Keywords: Visceral leishmaniasis; Leishmania infantum; Leishmania chagasi
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — Meglumine Antimoniate; amphotericin B, deoxycholate drug combination; Amphotericin B; liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Meglumine antimoniate (Active Comparator): Antimoniate of N-methylglucamine 20mg/kg/d, I.V. for 20 consecutive days.
  Interventions: Drug: Antimoniate of N-methylglucamine
- Liposomal Amphotericin B (Experimental): Liposomal amphotericin B 3mg/kg/d I.V. for 7 consecutive days.
  Interventions: Drug: Liposomal amphotericin B
- Amphotericin B (Experimental): Amphotericin B deoxycholate 1mg/kg/d I.V. for 14 consecutive days. This arm was suspended in September 19th, 2012, because of a relevant excess of adverse events and serious adverse events associated with this experimental intervention in comparison with the active comparator and the other two experimental arms. The suspension of this study arm was supported by a DSMB statement.
  Interventions: Drug: amphotericin B deoxycholate
- Combination therapy (Experimental): Liposomal amphotericin B 10mg/kg/d, I.V. single dose on day 0 plus Antimoniate of N-methylglucamine 20mg/kg/d for 10 consecutive days on days 1 to 10.
  Interventions: Drug: Liposomal amphotericin B; Drug: Antimoniate of N-methylglucamine

INTERVENTIONS:
Drug: Antimoniate of N-methylglucamine — Antimoniate of N-methyl glucamine 20mg/kg/d of pentavalent antimonial, I.V. for 20 consecutive days.
  Other Names: Glucantime
  Arms: Meglumine antimoniate
Drug: amphotericin B deoxycholate — 1mg/kg/d, I.V. for 14 consecutive days.
  Other Names: Fungizone; Anforicin B
  Arms: Amphotericin B
Drug: Liposomal amphotericin B — 3mg/kg/d, I.V. for 7 consecutive days.
  Other Names: AmBisome
  Arms: Liposomal Amphotericin B
Drug: Liposomal amphotericin B — 10mg/kg/d, I.V. single dose.
  Other Names: AmBisome
  Arms: Combination therapy
Drug: Antimoniate of N-methylglucamine — 20mg/kg/d of pentavalent antimonial I.V. for 10 days
  Other Names: Glucantime
  Arms: Combination therapy

SUMMARY:
This study is aimed to compare the efficacy and safety of medications currently used in Brazil for treatment of visceral leishmaniasis. The investigators will compare the effects of meglumine antimoniate, two formulations of amphotericin B: deoxycholate and liposomal, and a combination of meglumine plus the liposomal amphotericin B formulation. The study is designed to demonstrate the difference in efficacy measured as cure rate at six months after treatment and the safety profile based on the adverse event rate observed with each intervention.

DETAILED DESCRIPTION:
Visceral leishmaniasis is a relevant public health problem in Brazil with approximately 3500 cases registered every year. Eight percent lethality rate has been observed during the past decade in spite of free of charge availability of antileishmanial drugs supplied by the public health system.

The present study was designed as a phase IV, multicentric, open label, active controlled clinical trial targeted to visceral leishmaniasis adult and pediatric cases.

The current drugs approved for visceral leishmaniasis treatment in Brazil will be compared in four treatment groups: meglumine antimoniate, amphotericin B deoxycholate, liposomal amphotericin B and a combination of single dose of liposomal amphotericin B plus meglumine antimoniate. Meglumine antimoniate treated patients will constitute the active control group.

Drugs will be compared based on the cure rate observed after six months follow-up.

The study arm submitted to treatment with Amphotericin B deoxycholate was suspended in September 2012.

ELIGIBILITY:
Inclusion Criteria:

* patients with visceral leishmaniasis characterized by fever plus hepatomegaly or splenomegaly with at least one positive result in the following laboratory tests:
* direct observation of leishmania amastigotes in bone marrow smear
* leishmania in vitro culture from bone marrow aspirates
* leishmania kDNA amplification by PCR in bone marrow or peripheral blood samples
* rK39 immunochromatographic rapid test performed on serum sample

Exclusion Criteria:

* pregnancy
* HIV infection
* chronic diseases such as diabetes mellitus,kidney, liver or cardiac diseases, schistosomiasis, malaria or tuberculosis
* immune disorders or use of drugs which interferes with the immune response
* treatment with drugs with increased risk for toxicity associated with the study drugs
* exposure to antileishmanial drugs during the past six months
* I.V. drug users
* episodes of visceral leishmaniasis relapse
* hypersensibility to the study drugs
* difficulties for accomplishing the follow-up schedule
* any of the following clinical signs of laboratory abnormalities: hepatic encephalopathy, generalized edema, toxemic individuals, severe malnutrition, jaundice, abnormal serum creatinine, bilirubin, INR > 2,0, platelet count < 20000/mm3

Ages: 6 Months to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 378 (Actual)
Dates: Start 2011-02; Primary Completion 2014-10 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Cure rate | 6 month
  Complete remission of clinical signs and symptoms, three months after treatment plus normal hematological lab evaluation and no relapse at sixth month follow-up.

SECONDARY OUTCOMES:
Improvement rate | 30 days
  Fever disappearing, stable or improving hematological lab abnormalities plus any spleen size reduction.
Relapse rate | (6 months post treatment) After treatment until the sixth month of follow-up
  Reappearing of signs and symptoms after any improvement observed after treatment, during the six months follow-up period.
Serious adverse events rate | During (day one) and within the six months follow-up
  Rate of adverse events defined as conditions which fulfilled any of the following: results in death, is life threatening, requires inpatient hospitalization or prolongs hospitalization, results in persistent or significant disability/incapacity, causes a congenital anomaly or birth defect or it is considered as a important medical event for the responsible clinician.
Adverse event rate and intensity | During (day one) treatment and within the six months follow-up
  Cumulative rate of any adverse event, including clinical, laboratory and electrocardiographic abnormalities observed within the treatment and follow-up periods. All adverse events will be graded using an adapted ACTG 0-4 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos HN Costa, MD PhD, Principal Investigator — Federal University of Piaui; Dorcas L Costa, MD PhD, Principal Investigator — Federal University of Piaui; Ana LT Rabello, MD PhD, Principal Investigator — Centro de Pesquisas Rene Rachou - Fiocruz - Minas Gerais; Silvio FG de Carvalho, MD PhD, Principal Investigator — Montes Claros State University - Unimontes; Andrea L de Carvalho, MD, Principal Investigator — Hospital Infantil Joao Paulo II - FHEMIG; Roque P de Almeida, MD PhD, Principal Investigator — Federal University of Sergipe; Fabiana P Alves, MD PhD, Study Director — Drugs for Neglected Diseases; Gustavo AS Romero, MD PhD, Study Chair — University of Brasilia; Robério D Leite, MD, PhD, Principal Investigator — Hospital São José de Doenças Infecciosas, Secretaria de Saúde do Estado do Ceará.
Locations (5):
- Brazil (5):
  - Hospital Universitário da Universidade Federal de Sergipe, Sergipe, Aracaju
  - Hospital São José de Doenças Infecciosas, Fortaleza, Ceará
  - Hospital Infantil João Paulo II - FHEMIG, Belo Horizonte, Minas Gerais
  - Hospital Universitário Clemente de Faria - Universidade Estadual de Montes Claros, Montes Claros, Minas Gerais
  - Hospital de Doencas Infecto Contagiosas - HDIC, Teresina, Piauí

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Romero GAS, Costa DL, Costa CHN, de Almeida RP, de Melo EV, de Carvalho SFG, Rabello A, de Carvalho AL, Sousa AQ, Leite RD, Lima SS, Amaral TA, Alves FP, Rode J; Collaborative LVBrasil Group. Efficacy and safety of available treatments for visceral leishmaniasis in Brazil: A multicenter, randomized, open label trial. PLoS Negl Trop Dis. 2017 Jun 29;11(6):e0005706. doi: 10.1371/journal.pntd.0005706. eCollection 2017 Jun. PMID 28662034